CLINICAL TRIAL: NCT03591835
Title: Is Nasal Septum-tragus Length Safe in Neonatal Endotracheal Intubation?
Brief Title: Endotracheal Tube Placement in Neonatal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Associated Professor, M.D., Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TEP2018133
Record Dates: First submitted 2018-06-22; First posted 2018-07-19 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Neonatal Respiratory Failure
Keywords: Nasal septum-tragus length; newborn

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The radiologist who will determine endotracheal tube placement in the X-ray
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight+6 (Active Comparator): For the Tochen formula in Group 1, ETT depth will be calculated by taking the infant's actual weight within the last 24 h and adding 6 cm.
  Interventions: Other: Weight+6
- NTL+1 (Active Comparator): The infants in Group 2 will be intubated by measuring the NTL, the distance from the basement of the nasal septum to the the tragus of the ear.
  Interventions: Other: NTL+1

INTERVENTIONS:
Other: Weight+6 — For the Tochen formula in Group 1, ETT depth will be calculated by taking the infant's actual weight within the last 24 h and adding 6 cm.
  Arms: Weight+6
Other: NTL+1 — The infants in Group 2 will be intubated by measuring the NTL, the distance from the basement of the nasal septum to the the tragus of the ear. Measurements will be recorded as centimeters.
  Arms: NTL+1

SUMMARY:
Endotracheal intubation is a frequent procedure performed in neonates with respiratory distress. Clinicians use different methods to estimate the intubation insertion depth.

In this study, the investigators aimed to compare the two different methods (kilogram + 6 cm and nasal septum-tragus length (NTL) + 1 cm) used to determine the endotracheal intubation insertion depth.

DETAILED DESCRIPTION:
Endotracheal intubation is a frequent procedure performed in neonates with respiratory distress. The ideal location of the tube is between the top of the 1st thoracic vertebra and the bottom of the 2nd thoracic vertebra in the X-ray. Clinicians use different methods to estimate the intubation insertion depth.

In this study, investigators aimed to compare the two different methods (kilogram+6 cm and nasal septum-tragus length (NTL)+ 1 cm) used to determine the endotracheal intubation insertion depth.

In this multicentre randomized prospective study, infants who had intubation indications in neonatal intensive care unit will be enrolled. The intubation tube will be fixed at the lip level using the Tochen formula (Group 1) or the NTL+1 cm formula (Group 2). The same brand endotracheal tubes will be used and after intubation the chest radiograph will be performed in the neutral position. Chest X-ray will be evaluated blindly by a single radiologist in the digital environment (above T1, in place and below T2).

ELIGIBILITY:
Inclusion Criteria:.

* Infants who had intubation indications (cardiopulmonary failure, respiratory distress or surfactant administration) in the neonatal intensive care unit

Exclusion Criteria:

* Craniofacial, vertebral and genetic anomalies
* Those whose parents decline consent

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Correct placement of the ETT | Up to 1 hour
  After intubation a portable chest radiograph with digitalized measurements will be obtained to document ETT position. Head at the time of the radiograph will be stabilized in the neutral position. Chest X-ray will be evaluated blindly by a single radiologist in the digital environment (above upper border of T1, in place and below lower border of T2).

SECONDARY OUTCOMES:
Pneumothorax | Up to postmenstrual 52 weeks or till discharge
  Pneumothorax by transillumination confirmed by chest x-ray.
Bronchopulmonary displasia (BPD) | Postnatal age of 28 days or till discharge
  BPD will be defined according to National Institutes of Health criteria.
Mortality | Up to postmenstrual 52 weeks or till discharge
  We will record who died until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yekta Oncel, M.D., Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (5):
- Turkey (Türkiye) (5):
  - Zekai Tahir Burak Maternity Teaching Hospital, Ankara
  - Diyarbakır Gazi Yaşargil Training and Research Hospital, Diyarbakır
  - Ege University, Izmir
  - Izmir Tepecik Training and Research Hospital, Izmir
  - Şanlıurfa Training and Research Hospital, Sanliurfa

IPD SHARING:
Plan to Share IPD: Undecided